CLINICAL TRIAL: NCT00284128
Title: Double-blind, Randomized, Parallel-group, Dose Ranging, Multicenter Study to Evaluate the Efficacy and Safety of 2.5, 10, 35 and 50 mg AVE 7688 Once Daily, Using 100 mg Losartan-potassium Once Daily as Calibrator, for 12 Months Treatment, in Patients With Mild to Moderate Hypertension
Brief Title: AVE7688 in Patients With Mild to Moderate Blood Pressure
Acronym: RAVEL-1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI6032
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Hypertension
Keywords: Cardiovascular Disease C14; vascular disease C14.907; hypertension C14.907.489
MeSH Terms: conditions — Hypertension | interventions — AVE 7688; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- ilepatril (2.5 mg ) once daily (Experimental): AVE7688 oral administration
  Interventions: Drug: AVE7688
- ilepatril (10 mg) once daily (Experimental): AVE7688 oral administration
  Interventions: Drug: AVE7688
- ilepatril (35 mg) once daily (Experimental): AVE7688 oral administration
  Interventions: Drug: AVE7688
- ilepatril (50 mg) once daily (Experimental): AVE7688 oral administration
  Interventions: Drug: AVE7688
- Losartan-potassium (100 mg) once daily (Other): oral administration
  Interventions: Drug: Losartan-potassium

INTERVENTIONS:
Drug: AVE7688 — oral administration (capsules)
  Other Names: ilepatril
  Arms: ilepatril (10 mg) once daily; ilepatril (2.5 mg ) once daily; ilepatril (35 mg) once daily; ilepatril (50 mg) once daily
Drug: Losartan-potassium — oral administration (capsules)
  Arms: Losartan-potassium (100 mg) once daily

SUMMARY:
The primary objective is to assess the antihypertensive efficacy of 4 different AVE 7688 doses on the change from baseline in trough diastolic blood pressure at the end of week 12.

The secondary objectives are:

* To assess the antihypertensive efficacy of 4 different AVE 7688 doses on the change from baseline in trough systolic blood pressure at the end of week 12
* To compare the percentages of responders after 12 week of treatment
* To evaluate the long term safety and tolerability of AVE 7688 with particular attention to angioedema

DETAILED DESCRIPTION:
This study is a prospective multi-center, randomized, double-blind, active-controlled parallel-group, dose ranging study with 5 treatment groups (AVE7688 at 4 different dosages, and losartan-potassium 100 mg). There will be 3 study phases: placebo lead-in, treatment, and follow-up.

During the placebo lead-in phase (duration 3 to 4 weeks), patients will discontinue concomitant treatment with any antihypertensive or vasodilating agents and will receive single-blind placebo until randomization. Patients who meet the inclusion and exclusion criteria will be randomized to receive once-daily oral doses of either 2.5, 10, 35 or 50 mg AVE7688, or 100 mg losartan-potassium.

The treatment phase will consist of two parts: an efficacy evaluation period, with a 2 week titration period (from randomization to week 2, visit T1 to visit T3) up to 12 weeks, followed by a long-term safety evaluation period until the end of week 52. Antihypertensive treatment such as diuretics, beta blockers or calcium channel blockers can be introduced or re-introduced if indicated during the long term safety evaluation period but angiotensin converting enzyme inhibitors (ACE-I) or angiotensin receptor blockers (ARBs) are not permitted.

An additional visit (visit F1) will occur two weeks after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild-to-moderate, treated or untreated, essential hypertension, as defined by the JNC VII (Joint National Committee on the Prevention, Detection, Evaluation, and

Treatment of High Blood Pressure, Seventh report ) guidelines who meet the following BP eligibility criteria:

* mean SeSBP (Seated systolic blood pressure) ≥140 mm Hg and <180 mm Hg and mean SeDBP (Seated diastolic blood pressure) ≥90 mm Hg and <110 mm Hg at two consecutive qualifying visits in the placebo lead-in phase
* variability between the mean BP measurements on the 2 consecutive qualifying visits is less or equal 7 mm Hg for SeDBP.

Exclusion Criteria:

* Refusal or inability to give informed consent
* Patients who have previously been treated with AVE7688
* Patients who cannot stop their anti-hypertensive treatment
* Known history of secondary hypertension, including patients with endocrine disorders such as pheochromocytoma, active hyperthyroidism, or untreated hypothyroidism
* Severe hypertension
* Women of child bearing potential, who have a positive serum pregnancy test, or who do not agree to use an accepted method of contraception
* Women who are breast feeding
* Patients with non-cardiac progressive fatal disease
* Patients with immunological or hematological disorders
* Requirement for concomitant treatment that could bias the primary evaluation
* Unstable insulin-dependent diabetes mellitus
* History of stroke, intracranial hemorrhage or transitory ischemic attack within the previous year
* Likelihood of poor compliance both with treatment and study design
* Patient is the investigator, sub-investigator, research assistant, pharmacist, study coordinator, or other staff member or relative there of directly involved in the conduct of the study
* Administration of any investigational drug within the preceding 30 days
* Abuse of drugs or alcoholic beverages within 1 year prior to the start of the study
* Patients taking herbal or dietary compounds that have the potential to influence blood pressure
* Contraindications to losartan-potassium as per local package insert
* History of hypersensitivity or angioedema with ACE inhibitors or NEP inhibitors, patients with hereditary or idiopathic angioedema, patients with allergic reaction in which urticaria or angioedema was the manifestation
* Impaired hepatic function
* Known unilateral or bilateral renal artery stenosis
* Serum potassium > 5.5 mmol/L
* Impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1940 (Actual)
Dates: Start 2005-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough diastolic blood pressure at the end of week 12. | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in trough systolic blood pressure at the end of week 12, percentages of responders after 12 week of treatment. | 12 weeks
Evaluation of long term safety and tolerability of AVE7688 with particular attention to angioedema. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No